CLINICAL TRIAL: NCT05466812
Title: Efficacy Evaluation of Strontium-89 Chloride for Differentiated Thyroid Cancer With Bone Metastases
Brief Title: Efficacy of Sr-89 for Differentiated Thyroid Cancer With Bone Metastases
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Yansong Lin, Vice director, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZS-3477
Record Dates: First submitted 2022-07-12; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Thyroid Neoplasm Follicular; Bone Metastases
MeSH Terms: interventions — strontium chloride

STUDY DESIGN:
Intervention Model Description: Sr-89 treatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sr-89 treated group (Experimental): Sr-89 treatment
  Interventions: Drug: Sr-89

INTERVENTIONS:
Drug: Sr-89 — 1. strontium-89 chloride treatment
  2. periodical evaluation and follow-up
  Other Names: strontium-89 chloride

SUMMARY:
Using sensitive markers (such as thyroglobulin, etc) to evaluate the efficacy of strontium-89 chloride (Sr-89) in differentiated thyroid cancer with bone metastases with an aim to breaking out of its palliation effect for bone pain.

DETAILED DESCRIPTION:
Using biochemical markers (such as thyroglobulin), functional markers (such as change of tumor-background ratio on bone scan), etc to evaluate the efficacy of strontium-89 chloride (Sr-89) in differentiated thyroid cancer with bone metastases with an aim to breaking out of its palliation effect for bone pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients of differentiated thyroid cancer
* Positive uptake by bone metastases on bone scan
* Planing to have Sr-89 treatment

Exclusion Criteria:

* Having received treatment for bone metastases within one month of the study (such as radiotherapy, surgery, targeted therapy, chemotherapy, etc., among which denosumab and bisphosphate were allowed as basic treatment)
* Having received radioactive iodine therapy within half a year before the study
* There are bone related events, such as fracture, spinal cord compression, etc.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-13 (Estimated); Primary Completion 2024-07-13 (Estimated); Study Completion 2025-07-13 (Estimated)

PRIMARY OUTCOMES:
Change of serum thyroglobulin (Tg) level | Through study completion, an average of 1 week in the first months and 1 month thereafter, up to 6 months
  Change of serum Tg level
Change of serum thyroglobulin antibody (TgAb) level | Through study completion, an average of 1 week in the first months and 1 month thereafter, up to 6 months
  Change of serum TgAb level
Change of serum calcium level | Through study completion, an average of 1 week in the first months and 1 month thereafter, up to 6 months
  Change of serum calcium level
Change of serum alkaline phosphatase (ALP) level | Through study completion, an average of 1 week in the first months and 1 month thereafter, up to 6 months
  Change of ALP level
Change of tumor-background ratio on bone scan | Baseline, 3 months and 6 months
  Change from baseline tumor-background ratio on bone scan at 3 months and 6 months
Change of standardized uptake value (SUV) on positron emission tomography/ computed tomography (PET/CT) | Baseline, 3 months and 6 months
  Change from baseline SUV on PET/CT at 3 months and 6 months

SECONDARY OUTCOMES:
Structural change on image | Baseline, 3 months and 6 months
  Structural change on image at 3 months and 6 months
Numerical rating scale (NRS) for pain | Through study completion, an average of 1 week in the first months and 1 month thereafter, up to 6 months
  Scale of 0 to 10, 0=no pain, 10=worst imaginable pain
Skeletal related event (SRE) | Up to 6 months
  Any SRE such as pathological fractures, surgery/radiotherapy for pain/prevention of fractures, hypercalcemia, and spinal cord compression.
Analgesics | Up to 6 months
  Quantification of the use of analgesics and changes over time

CONTACTS AND LOCATIONS:
Overall Officials: Yan-Song Lin, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China